CLINICAL TRIAL: NCT04406129
Title: Effect of Fecal Microbiota Transplantation on Primary Hypertension and the Underlying Mechanism of Gut Microbiome Restoration: a Randomized Clinical Trial
Brief Title: Effect of Gut Microbiome Restoration on Primary Hypertension Via FMT
Acronym: FMT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Jun Cai, Professor, Director of Hypertension Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-GZ10 (Part I)
Record Dates: First submitted 2020-05-20; First posted 2020-05-28 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Hypertension
Keywords: Hypertension; Microbiome; Treatment; Fecal Microbiota Transplantation
MeSH Terms: conditions — Hypertension | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT capsules (Experimental): Intervention: FMT capsules containing extensively screened donor stool. FMT capsules will be orally taken on Day 1, Day 7 (Week 1) and Day 14 (Week 2).
  Interventions: Biological: FMT capsules
- Placebo capsules (Placebo Comparator): Intervention: Placebo capsules that do not contain donor stool or any active drug. Placebo capsules will be orally taken on Day 1, Day 7 (Week 1) and Day 14 (Week 2).
  Interventions: Other: Placebo capsules

INTERVENTIONS:
Biological: FMT capsules — Intervention: FMT capsules containing extensively screened donor stool.
  Arms: FMT capsules
Other: Placebo capsules — Intervention: Placebo capsules that do not contain donor stool or any active drug.
  Arms: Placebo capsules

SUMMARY:
Mounting preclinical and clinical evidences have proved the causal role of gut microbiota on the pathogenesis of primary hypertension. Restoration of gut microbiota ameliorated high BP in rodents and/or human cases.A hypothesis is thus raised that gut microbiome restoration can be a potential approach to ameliorate hypertension. This pilot study will utilize fecal microbiota transplantation (FMT) capsules, in comparison with placebo capsules, to investigate the effect, safety and underlying mechanisms of gut microbiome restoration on primary hypertension.

DETAILED DESCRIPTION:
Primary hypertension is a most prevalent cardiovascular diseases, and becomes a severe global public health issue because of the high morbidity and potential risk to other cardiovascular diseases. Several animal studies and diverse patient cohorts reported that the disorder of gut microbiome correlated with hypertension. Based on the investigators' previous work findings of metagenomics analysis, fecal transplantation and metabolomics changes in hypertension and pre-hypertension patients, a casual role of gut microbiome disorder was observed in primary hypertension and raised a hypothesis that gut microbiome restoration can be a potential approach to ameliorate hypertension. Recent studies indicated FMT, prebiotics, probiotics, dietary changes and other methodologies can assist gut microbiome restoration in diseases such as type 2 diabetes. The investigators therefore develop two pilot studies respectively utilizing FMT capsules (Pilot Study I) and innovative dietary changes (Pilot Study II) to explore the effect, safety and underlying mechanisms of gut microbiome restoration on hypertension. These pilot studies also present as the clinical translational section of the research project "The Role of Gut Microbiome in the Pathogenesis of Essential Hypertension"(Project ID 81630014, sponsored by National Natural Science Foundation of China).

This study is the Study I:

Objective: To explore the effect, safety and underlying mechanisms of gut microbiome restoration via FMT on primary hypertension.

Study Design: A multicenter, randomized, double-blinded, placebo-controlled pilot study.

Data quality control and statistical analysis: The investigators have invited professional statistic analysts to assist analyzing data and a third party to supervise data quality.

Ethics: The Ethics Committee of Fuwai Hospital approved this study. Informed consents before patient enrollment are required.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~60 years.
2. Established Diagnosis of Grade 1 Hypertension (initial diagnosis or free from antihypertensive drugs within a month): 140mmHg≤ Office SBP<160mmHg for three measurements at different days without any antihypertensive medications, according to the "2010 Chinese Guidelines for Prevention and Treatment of Hypertension".
3. Patients with informed consent after thorough explanation.

Exclusion Criteria:

1. Antibiotics or probiotics usage within last 4 weeks
2. Participants of other clinical trials related to hypertension currently or within last 3 months
3. Antihypertensive medications usage currently or within last month
4. Diagnosed secondary hypertension
5. Severe hepatic or renal diseases ((ALT >3 times the upper limit of normal value, or end stage renal disease on dialysis or eGFR <30 mL/min/1.73 m2, or serum creatinine >2.5 mg/dl [>221 μmol/L])
6. History of large atherosclerotic cerebral infarction or hemorrhagic stroke (not including lacunar infarction and transient ischemic attack [TIA])
7. Hospitalization for myocardial infarction within last 6 months; Coronary revascularization (PCI or CABG) within last 12 months; Planned for PCI or CABG in the next 12 months.
8. Sustained atrial fibrillation or arrhythmias at recruitment disturbing the electronic BP measurement.
9. NYHA class III-IV heart failure; Hospitalization for chronic heart failure exacerbation within last 6 months.
10. Severe valvular diseases; Potential for surgery or percutaneous valve replacement within the study period.
11. Dilated cardiomyopathy; Hypertrophic cardiomyopathy; Rheumatic heart disease; Congenital heart disease.
12. Other severe diseases influencing the entry or survival of participants, such as malignant tumor or acquired immune deficiency syndrome.
13. Cognitive impairment or severe neuropsychiatric comorbidities who are incapable of providing their own informed consent.
14. Participants preparing for or under pregnancy and/or lactation.
15. Other conditions inappropriate for recruitment according to the investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Change for Office Systolic Blood Pressure (SBP) | From baseline to Day 30
  Change for Office Systolic Blood Pressure (SBP)

SECONDARY OUTCOMES:
Change for Office SBP | Baseline, Day 7, Day 14, Day 30, Day 60, Day 90
  Change for Office SDBP
Change for Office Diastolic Blood Pressure (DBP) | Baseline, Day 7, Day 14, Day 30, Day 60, Day 90
  Change for Office Diastolic Blood Pressure (DBP)
Change for Home Systolic Blood Pressure (SBP) | Baseline, Day 7, Day 14, Day 30, Day 60, Day 90
  Change for Home Systolic Blood Pressure (SBP)
Change for Home Diastolic Blood Pressure (DBP) | Baseline, Day 7, Day 14, Day 30, Day 60, Day 90
  Change for Home Diastolic Blood Pressure (DBP)
Change for average SBP via 24-hour Ambulatory BP Monitoring | Baseline, Day 30, Day 90
  Change for average SBP via 24-hour Ambulatory BP Monitoring
Change for average DBP via 24-hour Ambulatory BP Monitoring | Baseline, Day 30, Day 90
  Change for average DBP via 24-hour Ambulatory BP Monitoring
Change for daytime average SBP via 24-hour Ambulatory BP Monitoring | Baseline, Day 30, Day 90
  Change for daytime average SBP via 24-hour Ambulatory BP Monitoring
Change for daytime average DBP via 24-hour Ambulatory BP Monitoring | Baseline, Day 30, Day 90
  Change for daytime average DBP via 24-hour Ambulatory BP Monitoring
Change for nightime average SBP via 24-hour Ambulatory BP Monitoring | Baseline, Day 30, Day 90
  Change for nightime average SBP via 24-hour Ambulatory BP Monitoring
Change for nightime average DBP via 24-hour Ambulatory BP Monitoring | Baseline, Day 30, Day 90
  Change for nightime average DBP via 24-hour Ambulatory BP Monitoring
Change for Ankle-Brachial Blood Pressure Index(ABI) | Baseline, Day 90
  Change for ABI as an objective measurement of arterial insufficiency based on the ratio of ankle systolic pressure to brachial systolic pressure.
Number of Participants with Adverse Events (AEs) as a Measure of Safety | All AEs over 3 months
  Number of Participants with Adverse Events (AEs) as a Measure of Safety
Changes in Intestinal Microbiota Composition Pre- and Post-intervention via Metagenomic Analysis | Baseline, Day 7, Day 14, Day 30, Day 60, Day 90
  Changes in Intestinal Microbiota Composition Pre- and Post-intervention (FMT or Placebo) via Metagenomic Analysis, stratified by:
  1. Randomisation
  2. Change in Office SBP
Changes in Intestinal Microbiota Function Pre- and Post-intervention via Metagenomic Analysis | Baseline, Day 7, Day 14, Day 30, Day 60, Day 90
  Changes in Intestinal Microbiota Function Pre- and Post-intervention (FMT or Placebo) via Metagenomic Analysis, stratified by:
  1. Randomisation
  2. Change in Office SBP
Durability of Engraftment of Donor Microbiome Following FMT | Baseline, Day 7, Day 14, Day 30, Day 60, Day 90
  Durability of engraftment of donor microbiome following FMT, measured by similarity comparison of intestinal microbiota composition between donor and recipient
Changes in Intestinal Metabolite Composition Pre- and Post-intervention via Metabolomic Analysis | Baseline, Day 7, Day 14, Day 30, Day 60, Day 90
  Changes in Intestinal Metabolite Composition Pre- and Post-intervention (FMT or Placebo) via Metabolomic Analysis, stratified by:
  1. Randomisation
  2. Change in Office SBP
Changes in Serum Metabolite Composition Pre- and Post-intervention via Metabolomic Analysis | Baseline, Day 7, Day 14, Day 30, Day 60, Day 90
  Changes in Serum Metabolite Composition Pre- and Post-intervention (FMT or Placebo) via Metabolomic Analysis, stratified by:
  1. Randomisation
  2. Change in Office SBP
Change for Fasting Blood Glucose Level | Baseline, Day 90
  Change for Fasting Blood Glucose Level
Change for Blood Lipid Level (Total Cholesterol, Total Triglyceride, Low Density Lipoprotein Cholesterol, High Density Lipoprotein Cholesterol) | Baseline, Day 90
  Change for Blood Lipid Level (Total Cholesterol, Total Triglyceride, Low Density Lipoprotein Cholesterol, High Density Lipoprotein Cholesterol)
Change for Body Mass Index | Baseline, Day 90
  Change for Body Mass Index

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cai, MD,PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (7):
- China (7):
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Shantou University, Shantou, Guangdong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Southern University of Science and Technology Hospital, Shenzhen, Shenzhen
  - The People's Hospital of Ji Xian District, Tianjin, Tianjin Municipality
  - Fuwai Yunnan Cardiovascular Hospital, Kunming, Yunnan

REFERENCES:
- [Background] Li J, Zhao F, Wang Y, Chen J, Tao J, Tian G, Wu S, Liu W, Cui Q, Geng B, Zhang W, Weldon R, Auguste K, Yang L, Liu X, Chen L, Yang X, Zhu B, Cai J. Gut microbiota dysbiosis contributes to the development of hypertension. Microbiome. 2017 Feb 1;5(1):14. doi: 10.1186/s40168-016-0222-x. PMID 28143587
- [Background] Cammarota G, Ianiro G, Tilg H, Rajilic-Stojanovic M, Kump P, Satokari R, Sokol H, Arkkila P, Pintus C, Hart A, Segal J, Aloi M, Masucci L, Molinaro A, Scaldaferri F, Gasbarrini G, Lopez-Sanroman A, Link A, de Groot P, de Vos WM, Hogenauer C, Malfertheiner P, Mattila E, Milosavljevic T, Nieuwdorp M, Sanguinetti M, Simren M, Gasbarrini A; European FMT Working Group. European consensus conference on faecal microbiota transplantation in clinical practice. Gut. 2017 Apr;66(4):569-580. doi: 10.1136/gutjnl-2016-313017. Epub 2017 Jan 13. PMID 28087657
- [Background] Translating Microbiome Research into Therapies: The Path Ahead. Cell. 2020 Apr 2;181(1):20-21. doi: 10.1016/j.cell.2020.03.009. No abstract available. PMID 32243790
- [Derived] Fan L, Chen J, Zhang Q, Ren J, Chen Y, Yang J, Wang L, Guo Z, Bu P, Zhu B, Zhao Y, Wang Y, Liu X, Wang W, Chen Z, Gao Q, Zheng L, Cai J. Fecal microbiota transplantation for hypertension: an exploratory, multicenter, randomized, blinded, placebo-controlled trial. Microbiome. 2025 May 23;13(1):133. doi: 10.1186/s40168-025-02118-6. PMID 40410854
- [Derived] Fan L, Ren J, Chen Y, Wang Y, Guo Z, Bu P, Yang J, Ma W, Zhu B, Zhao Y, Cai J. Effect of fecal microbiota transplantation on primary hypertension and the underlying mechanism of gut microbiome restoration: protocol of a randomized, blinded, placebo-controlled study. Trials. 2022 Feb 24;23(1):178. doi: 10.1186/s13063-022-06086-2. PMID 35209934